CLINICAL TRIAL: NCT04649593
Title: The Giving Birth Project, a Study of Labor Dystocia
Brief Title: The Study of Giving Birth, a Study About Treatment of Labor Dystocia
Acronym: GB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Eva Wiberg-Itzel, Associate professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GB1
Record Dates: First submitted 2020-11-22; First posted 2020-12-02 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Dystocia
MeSH Terms: conditions — Dystocia

STUDY DESIGN:
Intervention Model Description: According to the clinic's memo, when the labor is found to be dystocic, the woman is asked about her participation in the study. If the woman admits participation, she is included in the project. This is also noted in her journal.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- according to clinical guidlines (No Intervention): Dystocic progress and an observed low AFL value (< 12.0 mmol/l).
- intevention (Experimental): At dystocic labor and an observed high AFL value, the woman is randomized to one of the intended two study groups.
  Group 1) Delivery according to the clinic's guidelines in case labor dystocia, i.e., oxytocin stimulation Group 2) Two bags of Samarin mixed in a glass of water. After an hour, In case of lack of progress, oxytocin stimulation is started.
  Interventions: Dietary Supplement: Samarin

INTERVENTIONS:
Dietary Supplement: Samarin — Half of the group with a high AFL value will have a glass of Samarin to drink
  Arms: intevention

SUMMARY:
Labor dystocia is an intransigent, high-profile issue in obstetric care, which causes significant maternal morbidity in low resource settings and maternal dissatisfaction, and increased healthcare costs worldwide. Amniotic fluid lactate, (AFL), values have recently been shown to reflect the metabolic status of the uterus and high levels have a strong association with subsequent need for operative intervention due to dystocia. In sports medicine, it is known that lactic acid can affect muscular performance but be decreased by bicarbonate given orally before physical activity. Main Outcome Measures: If an intake of bicarbonate, one hour before stimulation with oxytocin in cases with a high AFL value, changes the AFL levels and enhances delivery outcome in dystocic deliveries.

Design: Randomized controlled trial

DETAILED DESCRIPTION:
Primary question: whether high AFL values (>12mmol/l) in women with observed dystocic labor are best treated by

1. to handle childbirth according to the clinic's current guidelines in case of labor dystocia, i.e. with oxytocin stimulation
2. an intake of bicarbonate (Samarin) dissolved in water given 1 hour before the oxytocin is started Primary outcome variable A comparison of the frequency of spontaneous vaginal delivery in the observed two described intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* dystocic labor with a need of oxytocin >=34w of gestation

Exclusion Criteria:

* Nondystocic labors.
* Women who don't understand Swedish or English
* Premature deliveries (<34w)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study is about labor. It means only women is the possible inclusion
Enrollment: 2000 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Labor outcome | through study completion, an average of 1 year
  Labor outcome in the different groups (spontaneous vaginal, VE or caesarean section)
AFL values | through study completion, an average of 1 year
  AFL-values to be at different times during labor

SECONDARY OUTCOMES:
The use of oxytocin | through study completion, an average of 1 year
  Oxytocin stimulation (number of hours of stimulation and amount of oxytocin given),

CONTACTS AND LOCATIONS:
Locations (1):
- Eva Wiberg-Itzel, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No